CLINICAL TRIAL: NCT06639776
Title: Sexual Functioning After Erection Prosthesis Placement in Post Phalloplasty Transgender Persons: a Retrospective Cohort
Brief Title: Sexual Functioning After Erection Prosthesis Placement in Post Phalloplasty Transgender Persons
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2023-0605
Record Dates: First submitted 2024-08-19; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Transgenderism; Erectile Dysfunction; Prosthesis Durability; Gender Dysphoria; Sexual Dysfunction
Keywords: Gender dysphoria; Transgender; Phalloplasty; Erectile dysfunction; Sexual function; Erection prosthesis; Penile epithesis; Medical device; Penile splint; Genital reconstruction; Patient Reported Outcome Measures (PROMs)
MeSH Terms: conditions — Transsexualism; Erectile Dysfunction; Prosthesis Failure; Gender Dysphoria; Sexual Dysfunction, Physiological | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Questionnaire — All erection prosthesis placements in post-phalloplasty transgender and gender non-conforming individuals at Ghent University Hospital from start of the gender clinic until June 2023 will be evaluated. All patients that are at least 6 months after erection prosthesis placement and currently have a functioning prosthesis in place are eligible and will be contacted. Upon inclusion and informed consent, the patient's medical files will be used to gather all necessary underlying medical information that is relevant to this study. will receive an email asking them to complete a questionnaire for themselves. At the end of this questionnaire the patient will be asked if they have a sexual partner and if this partner is willing to participate as well. After affirmation, the partner will be contacted in the same way.
  Patients will receive a series of questionnaires reviewing recent sexual activity, sexual preference, satisfaction with the erectile prosthesis and quality partner relationship.

SUMMARY:
This study aims to explore sexual satisfaction among transgender men and their partners following the placement of erectile prostheses after phalloplasty. While phalloplasty can create a neophallus, the lack of natural erectile tissue often necessitates the use of erectile aids, including internal prostheses. However, these prostheses, originally designed for cisgender men, face challenges when used in transgender patients, such as higher risks of complications, infections, and mechanical failures. Despite these issues, some studies report high patient satisfaction, though partner satisfaction rates are significantly lower. The study will use validated and non-validated questionnaires to assess satisfaction with various types of erectile prostheses, addressing the gap in understanding how these devices impact the sexual and relational functioning of both transgender men and their partners. These questionnaires will be provided to all included patients that are minimum 6 months after placement of an internal erection prosthesis and have a functional erection prosthesis in place

DETAILED DESCRIPTION:
Gender dysphoria is defined as a discomfort or dissatisfaction because of a discordance between the individual's assigned sex and their gender identity. A national survey of transgender adults in the United States has shown that 39% of their respondents experience psychological distress, which is eight times the rate in the United States population. Transition-related treatment contains counseling, psychotherapy, hormone therapy and gender-affirming surgery depending on what the individual desires. Gender-affirming surgery aims to change an individual's physical characteristics concordant with their gender identity and results in a reduction of psychological distress.

A part of this population will eventually undergo genital gender affirming surgery (GGAS) to align the appearance of the external genitalia as well. In transgender men, GGAS can be performed as metoidioplasty or phalloplasty with or without the removal of the native external genitalia. In metoidioplasty, the goal is to create anatomically looking but undersized external genitalia in which the clitoris forms the base of a micro-penis. In phalloplasty, anatomically sized external genitalia (phallus with or without urethra, scrotum, and perineum) are created using on the one hand a donor skin flap and on the other hand tissues from the original genitals. As there is no erectile tissue present in the neophallus after phalloplasty, it is usually not possible to penetrate a sexual partner without the use of external or internal erectile aids. In patients having undergone phalloplasty, a multitude of methods for obtaining phallic rigidity are available. One option can be the implantation of an internal erectile prosthesis.

Most types of erectile prostheses used in the transgender community have originally been designed for cisgender men. However, implanting such a prosthesis in the neophallus presents a number of challenges due to the differences with the anatomy of a native penis. As there are no cavernosal bodies with surrounding tunica albuginea that can be used as scaffold for anchoring of the prosthesis to the pubic bone there is an increased risk for distal extrusion, malposition and extensive mobility during use. Furthermore, vascularization of the neophallus is largely dependent on the one or two vessels supplying the flap(s), resulting in relative hypovascularization, delayed healing and an increased risk of infection. Finally, these types of prosthesis were originally made for an older population with erectile dysfunction. Most transgender patients are younger and sexually more active which could lead to mechanical failure of the erectile prosthesis; hence the life expectancy of implants is significantly reduced in this population. Consequently, penile implant surgery is associated with higher complications in a transgender population than in a cisgender population. The revision rate or explantation rate within 4 years follow-up ranges from 37.6% to 44% in several studies. Falcone et al. reported that up to 22% of the prostheses was explanted within 20 months. Within this study the patient and partner satisfaction were surveyed with a non-validated questionnaire. Up to 88% of patients were completely satisfied with the outcome of the phalloplasty and the erectile prosthesis, despite a significant complication rate. However, the partner satisfaction rate is significantly lower and rated at 60%. Without further discussion, Falcone et al. stated that his result should be explored in the future.

Recently, the Swiss company Zephyr Surgical Implants created the ZSITM 475 female-to-male (FTM) (Switzerland, Europe), the first erectile prosthesis specifically designed for transgender men after phalloplasty surgery. It contains several functions such as a large base plate for pubic bone fixation, a glans shaped tip, and a testicle-shaped pump, that have been conceived to answer several of the difficulties of prosthesis implantation. Recent publications on this prosthesis continue to report high complication rates. Verla et al. reported postoperative complications in 32% of the patients. Moreover, 23% of the devices were explanted within 18 months follow-up due to distal cylinder protrusion, infection, malpositioning, mechanical failure and urinary retention. In the paper of Neuville et al., the overall revision rate was 19% with a mean follow-up of 8.9 months, resulting from infection, mechanical failure and malpositioning. However, 92.8% of patients reported to be either satisfied or very satisfied with the erectile prosthesis and a mean EDITS score of 82 of 100.

To date, it is not possible to state which prosthesis is performing better in terms of complications and sexual satisfaction. A more comprehensive questionnaire is needed to understand the reported satisfaction of the patient according to the different types of prosthesis. As observed in the publication of Falcone et al., the low partner satisfaction rate should be explored further as this may impact patients' and partners' relational functioning. The current study aims to explore in more detail the sexual satisfaction in both transgender patients and their partners regarding erectile prosthesis placement using validated and non-validated questionnaires. These questionnaires will be provided to all included patients that are minimum 6 months after placement of an internal erection prosthesis and have a functional erection prosthesis in place

ELIGIBILITY:
Inclusion Criteria:

* Patient and partner age ≥ 18 years.
* Transgender or gender non-conforming individuals diagnosed according to the DSM-5 diagnostic criteria for gender dysphoria.
* Patients have undergone phalloplasty as a form of genital gender affirming surgery (any type of flap combination or technique is allowed).
* Erection prosthesis placement ≥ 6 months after phalloplasty, performed at the Ghent University Hospital. Any type of prosthesis is allowed.
* Patient has a functional erectile prosthesis at the time of the study. Number of erectile prosthesis is not relevant for inclusion.
* Patient is Dutch, English or French speaking.
* Voluntary signed and written consent by patient and their optional partner.

Exclusion Criteria:

* Patient age < 18 years.
* Cisgender patients treated with phalloplasty and/or erection prosthesis for various reasons.
* The erection prosthesis has been explanted or the current prosthesis is nonfunctional at time of data assessment.
* Erection prosthesis placement < 6 months before study start will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-phalloplasty transgender patients that have undergone erectile prosthesis placement at the Ghent University Hospital at least six months ago and in whom the erection prosthesis in place in functioning.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Treatment satisfaction | One-time questionnaire at least 6 months after erection prosthesis placement
  Assessed using the Erectile Dysfunction Inventory of Treatment Satisfaction questionnaire (EDITS)
  The EDITS provides two summative scores of 0-44 and 0-20 for patient and partner scores respectively. A higher score indicates a better treatment satisfaction. Higher scores indicate better outcome.
  With this questionnaire a number of subgroup analyses will be conducted. The obtained scores for treatment satisfaction for different types of erectile prostheses will be compared. Besides that, the difference in scores between patients and their partners will be explored. Another possible subgroup analysis will compare patients with different number of erectile prostheses placed.
  It was decided not to use a specific question from the EDITS patient questionnaire. It applies to the participant's erectile dysfunction which is not relevant to this study. The maximum score will therefore be 40.
Capability of vaginal and/or anal penetration of the participant and sexual functioning | One-time questionnaire at least 6 months after erection prosthesis placement
  Separate questions regarding penetration, sexual functioning and the experience of the patient and their optional partner are listed in the appendix for patient and their optional partner.
  Capability will be defined as full repetitive anal and/or vaginal penetration of the partner while using the prosthesis, which was not possible before implantation, without pain to patient and/or partner, until the end of the intended sexual intercourse.
  If penetration is not possible, the reasons for this incapacity will be noted.
  Patient and their optional partner indicate how desirable and/ or painful penetration was using a Likert slider question on a scale of 1 to 5.

SECONDARY OUTCOMES:
Relationship satisfaction, sexual satisfaction, and quality of life | One-time questionnaire at least 6 months after erection prosthesis placement
  Assessed using the Maudsley Marital Questionnaire (MMQ).
  The MMQ provides three summative scores of 0-80, 0-40 and 0-40 on relationship satisfaction, sexual satisfaction, and overall quality of life. Lower scores indicate better outcome.
  Only if the participant has a stable sexual relationship, the questionnaire will be filled out.
Patient willing to undergo redo surgery and recommendation to other patients | One-time questionnaire at least 6 months after erection prosthesis placement
  Assessed using separate Yes/No questions
• Use of previous external devices or aids before placement of an erectile prosthesis | One-time questionnaire at least 6 months after erection prosthesis placement
  Specific questions regarding previous devices or aids other than erectile prostheses are listed in the appendix for patient and their optional partner.
  Patient and their optional partner indicate how desirable penetration was with other aids using a Likert slider question on a scale of 1 to 5. This answer will be compared to the slider question regarding the capability of penetration with an erectile prosthesis.
Lower urinary tract symptoms (LUTS) and their impact on quality of life. | One-time questionnaire at least 6 months after erection prosthesis placement
  Assessed using the International Consultation on Incontinence Questionnaire - Male Lower Urinary Tract Symptoms (ICIQ-MLUTS)
  The ICIQ-MLUTS module, consisting of 13 questions, provides a summative score between 0 (asymptomatic) and 52 (most symptomatic).
  With this questionnaire, the severity of the lower urinary tract symptoms will be explored. These scores could possibly be correlated with the patient's satisfaction score, the urinary function and the prosthesis related complications.
Prosthesis related complications. | One-time questionnaire at least 6 months after erection prosthesis placement
  Prosthesis related complications are extracted from medical files. These will be correlated with the patients satisfaction score from the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Françoise Spinoit, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Department of Urology, University Hospital Ghent, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No